CLINICAL TRIAL: NCT07135856
Title: Comparative Analysis of Minimally Invasive and Open Sleeve Lobectomy Following Neoadjuvant Therapy in NSCLC: A Multicenter Retrospective Evaluation of Surgical Outcomes
Brief Title: Sleeve Lobectomy Following Neoadjuvant Therapy in NSCLC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); University of Padova, Padova, Italy (Unknown)
Responsible Party: Principal Investigator, Xinghua Cheng, Director, Head of Oncology Surgery, Clinical Professor, Shanghai Chest Hospital
Other Study IDs: ShanghaiChestNeoSleeve
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracotomy sleeve lobectomy: Patients who underwent open sleeve lobectomy following neoadjuvant therapy
- MIS sleeve lobectomy: Patients who underwent minimally invasive (i.e. VATS and RATS) sleeve lobectomy following neoadjuvant therapy

SUMMARY:
The goal of this observational, retrospective, multicenter cohort study is to evaluate the surgical and oncologic outcomes of sleeve lobectomy performed via minimally invasive (RATS/VATS) or open thoracotomy approaches in patients with non-small cell lung cancer (NSCLC) who have undergone neoadjuvant therapy, including chemotherapy, immunotherapy, or combination regimens. The main questions this study aims to answer are:

* Does minimally invasive sleeve lobectomy result in comparable or improved perioperative and postoperative outcomes compared to open thoracotomy following neoadjuvant treatment in NSCLC?
* Does surgical approach influence oncologic endpoints such as margin status, lymph node dissection, recurrence-free survival, and overall survival? This research addresses a critical gap in the thoracic oncology field by evaluating the safety, complexity, and efficacy of advanced surgical techniques in the context of evolving multimodal therapy paradigm. Findings may inform clinical decision-making and optimize patient selection in an era of increasing use of neoadjuvant strategies for resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed NSCLC
* Undergoing sleeve lobectomy with curative intent
* Receipt of neoadjuvant therapy (chemotherapy, immunotherapy, target therapy, etc.)
* Surgical approach: either minimally invasive (VATS or RATS) or open thoracotomy
* Availability of complete perioperative and follow-up data (minimum 12-month follow-up or until death)
* Signed informative consent

Exclusion Criteria:

* Sublobar resections (e.g., segmentectomy) or pneumonectomy
* Absence of neoadjuvant therapy
* Purely diagnostic surgical procedures
* Incomplete medical records or lost to follow-up
* Metastatic (stage IV) disease at time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve multiple thoracic surgery centers with experience in advanced surgical techniques for lung cancer, including sleeve resections and neoadjuvant management. Each center will contribute anonymized data from eligible cases, in accordance with local ethical approvals and data protection regulations.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
3-year RFS | 3 years
  In this study, the investigators will focus on the 3-year recurrence-free survival (RFS) of the participants between the two groups (open vs. MIS) for the comparison of the long-term oncologic outcomes, as the primary outcome.

SECONDARY OUTCOMES:
3-year OS | 3 years
  The investigators will also focus on the 3-year overall survival (OS) of the participants between the two groups (open vs. MIS) for the comparison of the long-term oncologic outcomes, as the secondary outcome.

OTHER OUTCOMES:
Intraoperative bleeding | up to 90 days
  The intraoperative bleeding will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes, measured in milliliter (mL).
Surgery duration | up to 90 days
  The surgery duration will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes, measured in minute (min).
Postoperative hospital stay | up to 90 days
  The postoperative hospital stay will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes, measured in day.
Postoperative complications | up to 90 days
  The postoperative complications will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes, showed in the number of the participants who occurred postoperative complications (n).
Perioperative mortality | up to 90 days
  The perioperative mortality will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes, showed in the number of the participants who died within 90 days of surgery (n).
Number of dissected lymph nodes | up to 90 days
  The number of dissected lymph nodes will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes (n).
Number of dissected lymph node stations | up to 90 days
  The number of dissected lymph node stations will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes (n).
Margin status | up to 90 days
  The margin status will be investigated between open versus MIS sleeve lobectomy as one of the perioperative outcomes, showed in the number of the participants who had the positive or negative surgical margins (n).
Postoperative ICU Length of Stay | up to 90 days
  The postoperative ICU length stay will be investigating between open versus MlS sleeve lobectomy as one of the perioperative outcomes, measured in days. If no ICU admission occurs, length of stay is recorded as 0 days.
Postoperative chest tube drainage duration | up to 90 days
  The postoperative chest tube drainage duration will be investigating between open versus MlS sleeve lobectomy as one of the perioperative outcomes, measured in days.
Postoperative pain scores | up to 90 days
  The postoperative pain scale will be investigating between open versus MlS sleeve lobectomy as one of the perioperative outcomes, measured with the Numeric Rating Scale (0-10) on postoperative days 1 and 2, and highest score during hospitalization.
Conversion rate to Thoracotomy | at surgery
  The conversion rate from minimally invasive (VATS or RATS) cases to open thoracotomy will be showed in numbers.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China